CLINICAL TRIAL: NCT01733576
Title: Enhancing Verbal Learning and Memory Using High-Definition Transcranial Direct Current Stimulation (HD-tDCS)
Brief Title: High-definition Transcranial Direct Current Stimulation (HD-tDCS) Verbal Learning
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Melissa Pigot, Research Assistant, The University of New South Wales
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CB64
Record Dates: First submitted 2012-11-26; First posted 2012-11-27 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Verbal Learning and Memory

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sham HD-tDCS (Sham Comparator)
  Interventions: Device: HD-tDCS
- Active HD-tDCS 1 (Active Comparator)
  Interventions: Device: HD-tDCS
- Active HD-tDCS 2 (Active Comparator)
  Interventions: Device: HD-tDCS
- Active HD-tDCS 3 (Active Comparator)
  Interventions: Device: HD-tDCS

INTERVENTIONS:
Device: HD-tDCS

SUMMARY:
This project will use a new form of non-invasive brain stimulation called high-definition transcranial direct current stimulation (HD-tDCS) to facilitate verbal learning. This form of stimulation is similar to transcranial direct current stimulation (tDCS) but allows for more spatially focused stimulation. We hypothesise that HD-tDCS when applied to regions of the brain important for learning and memory will improve verbal learning and memory compared to sham HD-tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 40 years
* Right-handed

Exclusion Criteria:

* concurrent medication likely to affect mental performance
* current history of drug or alcohol abuse or dependence
* any psychiatric or neurological disorder, recent head injury, or history of seizure or stroke.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Ray Auditory Verbal Learning Test (RAVLT)

CONTACTS AND LOCATIONS:
Locations (1):
- Black Dog Institute, Sydney, New South Wales, Australia